CLINICAL TRIAL: NCT03092076
Title: The Impact of Genotype on Pharmacokinetics and Antiplatelet Effects of Ticagrelor in Healthy Chinese
Acronym: IGPPT
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Guangdong Provincial People's Hospital (Other)
Responsible Party: Principal Investigator, ShiLong Zhong, Professor, Guangdong Provincial People's Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: GDREC2015143H(R1)
Record Dates: First submitted 2017-03-09; First posted 2017-03-27 (Actual); Last update posted 2017-03-27 (Actual); Status verified 2017-03

CONDITIONS: Healthy
Keywords: pharmacokinetics; antiplatelet effects; single nucleotide polymorphism (SNP)
MeSH Terms: interventions — Ticagrelor; ChAdOx1 nCoV-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Pharmacokinetics (Experimental): The pharmacokinetics characteristic of ticagrelor in healthy Chinese is investigated to provide the basis for its efficacy and safety of clinical treatment.
  Interventions: Drug: Ticagrelor
- Antiplatelet effects (Experimental): The antiplatelet effects of ticagrelor in healthy Chinese is investigated to provide the basis for its efficacy and safety of clinical treatment.
  Interventions: Drug: Ticagrelor
- The impact of genotype (No Intervention): The recovery time of platelet function following the administration of ticagrelor is widely varied that genetic variants maybe an underlying factor.The impact of genotype on pharmacokinetic parameters and ADP of ticagrelor is compared among different genotypes.

INTERVENTIONS:
Drug: Ticagrelor — 180 mg loading dose
  Other Names: Brilinta; AstraZeneca
  Arms: Antiplatelet effects; Pharmacokinetics

SUMMARY:
This study is a open and single center clinical trial in healthy Chinese.The objective of the study is to clarify the pharmacokinetics characteristics and antiplatelet effects of ticagrelor in Chinese and to investigate the impact of genotype.

DETAILED DESCRIPTION:
This is an open-label, single-does, nonrandomized study of ticagrelor in healthy volunteers carried out at a single center. Written informed consent will be obtained from all volunteers before initiation of the study. The study is approved by the Research Ethic Committee of Guangdong General Hospital. Fifty-one healthy Chinese will be recruited.

Venous blood will be collected at 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24 and 48h after taking 180mg ticagrelor orally. Urine collection intervals are at predose and 0 to 2, 2 to 4, 4 to 6, 6 to 9, 9 to 12, 12 to 16 and 16 to 24h after dosing. The concentration of ticagrelor and its metabolites will be analyzed using a separately validated liquid chromatography technique with tandem mass spectrometric detection (LC-MS/MS).

Besides，the basic principle of population pharmacodynamics(PPD) is applied to evaluate antiplatelet effects. Adenosine diphosphate(ADP)-stimulated platelet aggregation will be assessed at baseline, and 0.5h/1h, 2h, 4h/8h/24h, 48h/3d/5d and 7d after dosing.

The effects of genetic variants on antiplatelet and pharmacokinetic response to ticagrelor are investigated through a genome-wide association study (GWAS).

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18 - 45 years;
2. Sex: male and female;
3. Ethnicity: Chinese;
4. Good health as evidenced by the results of physical examination, vitals signs, electrocardiogram, and clinical laboratory test results, but there were exceptions if an abnormal value was considered not to be clinical significance;
5. Written informed consent.

Exclusion Criteria:

1. Any conditions known to interfere with the absorption, distribution, metabolism or excretion of drugs;
2. Intolerance or hypersensitivity to drugs whose mechanism is similar to that of ticagrelor;
3. Any history of taking medicines within half a month before enrollment;
4. Any history of whole blood transfusion within 2 months, blood elements transfusion or blood donation within 1 months before enrollment;
5. Participation in a clinical study within 3 months before enrollment;
6. Abuse of caffeine (> 5 units/day), alcohol(> 21 units /week), smoking(> 10 cigarettes/day);
7. Positive serology for Hbs antigen and HIV;
8. History of coagulation disorders.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 51 (Actual)
Dates: Start 2015-05-20 (Actual); Primary Completion 2015-10-24 (Actual); Study Completion 2016-06-16 (Actual)

PRIMARY OUTCOMES:
Genome-wide genotyping in 51 healthy Chinese | 10 weeks
  A total of 900,015 SNPs in a GWAS scan were genotyped with the Illumina HumanOmniZhongHua-8 BeadChip according to the protocol from Illumina. Prior to association analysis, a systematic quality control (QC) procedure was applied to the raw genotyping data to filter unqualified SNPs and samples. The effects of genetic variants on antiplatelet and pharmacokinetic response to ticagrelor are investigated through a genome-wide association study（GWAS）in 51 healthy Chinese .

SECONDARY OUTCOMES:
ADP-stimulated platelet aggregation | 8 weeks
  For platelet function tests, ADP-stimulated platelet aggregation was measured in ethylenediaminetetraacetic acid (EDTA) anticoagulated whole blood samples (2 x 2 mL) within 2 h of sampling using a Chrono-log Platelet Aggregation Systems. The platelet aggregation (PA) postdose till recovery to baseline was measured by light transmission method using ADP (20 μmol/L final concentration), and expressed as percentages. Since a sparse sampling design for platelet function testing was used, the missing platelet aggregation data during the recovery of platelet function were imputed using Bayesian simulation method. The time recovering 50% of maximum drug effect (RT50) were estimated individually, which were used to represent the antiplatelet effect.
Peak plasma concentration (Cmax) | 10 weeks
  A LC-MS/MS assay was developed and validated for simultaneous determination of ticagrelor, its metabolites, and internal standard (ferulic acid) in human plasma. Plasma samples were extracted with ethyl acetate. Peak plasma concentration (Cmax) of ticagrelor and M8 were estimated for each subject, using the non-compartmental analysis function in Phoenix WinNonlin software, version 6.3.
Time to peak plasma concentration (tmax) | 10 weeks
  A LC-MS/MS assay was developed and validated for simultaneous determination of ticagrelor, its metabolites, and internal standard (ferulic acid) in human plasma. Plasma samples were extracted with ethyl acetate. Time to peak plasma concentration (tmax) of ticagrelor and M8 were estimated for each subject, using the non-compartmental analysis function in Phoenix WinNonlin software, version 6.3.
Area under the plasma concentration-time curve (AUC) | 10 weeks
  A LC-MS/MS assay was developed and validated for simultaneous determination of ticagrelor, its metabolites, and internal standard (ferulic acid) in human plasma. Plasma samples were extracted with ethyl acetate. Area under the plasma concentration-time curve (AUC) of ticagrelor and M8 were estimated for each subject, using the non-compartmental analysis function in Phoenix WinNonlin software, version 6.3.
Accumulated amount of ticagrelor and its metabolites in urine | 10 weeks
  A LC-MS/MS assay was developed and validated for simultaneous determination of ticagrelor, its metabolites, and internal standard (gliclazide) in human urine. Urine samples were precipitated with 50% methanol/acetonitrile. Accumulated amount of ticagrelor and its metabolites in urine over 24 h was calculated. The relative accumulated amount was the product of the relative index and the urine volume (Compound/IS x Vurine).

CONTACTS AND LOCATIONS:
Overall Officials: Shilong Zhong, Ph.D, Principal Investigator — Guangdong Provincial People's Hospital

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Chen J, Xu G, Xie Z, Xie S, Luo W, Zhong S, Lai W. GPD2 inhibition impairs coagulation function via ROS/NF-kappaB/P2Y12 pathway. Cell Mol Biol Lett. 2025 Jul 18;30(1):84. doi: 10.1186/s11658-025-00759-x. PMID 40682019
- [Derived] Xu G, Liu JE, Liu X, Zhong W, Wang Z, Li H, Xiao X, Chen J, Zhong S, Lai W. DNA methylation mediates the genetic variants on ticagrelor major metabolite elimination and platelet function recovery after ticagrelor discontinuation. Epigenomics. 2022 May;14(10):601-613. doi: 10.2217/epi-2021-0461. Epub 2022 May 16. PMID 35574651
- [Derived] Zhu Q, Zhong W, Wang X, Mai L, He G, Chen J, Tang L, Liu S, Lai W, Zhong S. Pharmacokinetic and Pharmacogenetic Factors Contributing to Platelet Function Recovery After Single Dose of Ticagrelor in Healthy Subjects. Front Pharmacol. 2019 Mar 18;10:209. doi: 10.3389/fphar.2019.00209. eCollection 2019. PMID 30936830